CLINICAL TRIAL: NCT07026032
Title: Effects of Biofeedback Exercises on Severity of Dysphagia in Parkinson's Clients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01763 Gulalai Shafiq Khan
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Oropharyngeal Dysphagia
Keywords: Parkinson
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Two groups will be made. Group A and Group B. One group will have traditional exercises and the other will have exercises using the Biofeedback.
Who Masked: Participant
Masking Description: The participant will not be aware of the treatment protocol used for their comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Parkinson with dysphagia (Experimental): Diagnosed cases of Parkinson's disease having oropharyngeal dysphagia were taken. The experimental group received exercises through biofeedback.
  Interventions: Other: Biofeedback tool
- Parkinson with Dysphagia (Other): The second group, that was the control group received traditional tongue exercises.
  Interventions: Other: Biofeedback tool; Other: traditional exercises

INTERVENTIONS:
Other: Biofeedback tool — Biofeedback tool (tongueometer) will be used for experimental group, where as for control group the intervention used in traditional exercises.
Other: traditional exercises — traditional exercises were used for the control group

SUMMARY:
A randomized control trial will be conducted to test if there will be a significant effect or not, of biofeedback exercises vs traditional exercises for clients with oropharyngeal dysphagia in Parkinson's disease. For this purpose, 32 participants will be taken for the study. Half will be given traditional exercises where as the other half will be given exercises using the biofeedback; tongueomter.

DETAILED DESCRIPTION:
An RCT will be conducted on 32 Parkinson's patients having oropharyngeal dysphagia. FOIS and biofeedback will be used as a baseline instrument to determine the tongue strength and severity of dysphagia at the initial level of the study. The experimental group will perform tongue isometric pressure exercises using biofeedback for twelve sessions, four sessions per week. The control group will perform only traditional tongue-strengthening exercises for twelve sessions, four sessions per week. Both groups will receive therapy for 30 minutes. Both groups will undergo twelve sessions of exercises, starting after a baseline evaluation. Each patient will receive therapy for 30 minutes and have four sessions of therapy weekly. Two exercise protocols will be used. Protocol A will involve biofeedback strengthening exercises using the tongueometer. Protocol B will involve traditional tongue exercises to improve coordination and strength in tongue movement. The experimental group will be instructed to perform Protocol A while the control group will be instructed to perform Protocol B. Each group after randomization will undergo twelve sessions of exercises and baseline assessment will be taken at initial, middle, and final levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of Parkinson disease
* Diagnosed patients of oropharyngeal dysphagia with both genders

Exclusion Criteria:

* Cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
FOIS | 3 Weeks
  FOIS is a clinical tool used to assess the functional oral intake of food and liquids in patients with dysphagia. It is a 7-point observer rating clinical scale that was developed to document changes in functional oral intake of liquid and food in stroke patients. FOIS was used for baseline evaluation and post assessment of Experimental and Control group.
  The experimental group demonstrated a notable increase in FOIS scores, improving from 4 ± 1 at baseline to 6 ± 0 at post-assessment. This indicates significant improvements in swallowing behavior associated with the biofeedback method.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Nadir, Study Director — Riphah International University
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No